CLINICAL TRIAL: NCT02337816
Title: Role of Metabolomics in the Diagnosis of Endometriosis
Status: Completed | Type: Observational
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Other Study IDs: ENDOMETAB01
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Endometriosis
Keywords: Endometriosis; Metabolomics
MeSH Terms: conditions — Endometriosis | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine samples, blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis: Patients will undergo laparoscopic surgery in order to treat endometriosis. Biopsies will be performed for histological confirmation of the disease. Samples of urine and blood, with the purpose to study metabolitis, will be collected before surgery.
  Interventions: Procedure: laparoscopic surgery, obtainment of biological samples
- Controls: Patients will undergo laparoscopic surgery in order to treat benign gynecological diseases. Biopsies will be performed for histological confirmation of the disease. Samples of urine and blood,with the purpose to study metabolitis, will be collected before surgery.
  Interventions: Procedure: laparoscopic surgery, obtainment of biological samples

INTERVENTIONS:
Procedure: laparoscopic surgery, obtainment of biological samples

SUMMARY:
Endometriosis is one of the most common benign gynecological, affecting about 10% of premenopausal women. The pathophysiology of this disease is still not completely clear. Despite its prevalence, there is no blood test available for the diagnosis of endometriosis and the average delay time to diagnosis is 9.4 years.

Metabolomics is a scientific discipline that studies changes in metabolites related to the pathophysiology of the disease.

Aim of the study is to identify an alteration in the expression of the metabolites in women with endometriosis

ELIGIBILITY:
Inclusion Criteria:

* women of childbearing age ;
* written consent to laparoscopic surgery;
* written consent to the study .

Exclusion Criteria:

* Suspicion or diagnosis of malignant disease
* Inability or unwillingness to provide written consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women of childbearing age , patients of the University Hospital , suffering from benign gynecological disease
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Plasma and urine concentration of metabolites | At least one month after discontinuation of hormonal therapies , before laparoscopic surgery

REFERENCES:
- [Derived] Murgia F, Angioni S, D'Alterio MN, Pirarba S, Noto A, Santoru ML, Tronci L, Fanos V, Atzori L, Congiu F. Metabolic Profile of Patients with Severe Endometriosis: a Prospective Experimental Study. Reprod Sci. 2021 Mar;28(3):728-735. doi: 10.1007/s43032-020-00370-9. Epub 2020 Nov 10. PMID 33174185